CLINICAL TRIAL: NCT04516629
Title: Using the Objective Physiological Parameters to Test TCM Syndrome in Sub-health Subjects
Status: Completed | Type: Observational
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Other Study IDs: YM105101E
Record Dates: First submitted 2020-03-18; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2018-10

CONDITIONS: Health Status
Keywords: subhealth; obese; hypertension; sleep apnea syndrome; fatigue; TCM syndrome; physiological signal monitor system
MeSH Terms: conditions — Obesity; Hypertension; Sleep Apnea Syndromes; Fatigue

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: subjects with sub-health status
  Interventions: Diagnostic Test: heart rate variability, pulse diagnosis device

INTERVENTIONS:
Diagnostic Test: heart rate variability, pulse diagnosis device — check heart rate and pulse rate

SUMMARY:
Background: Suboptimal health status (SHS) is a dynamic state potential clinical stage or prior psychosomatic disease stage during which people have not been diagnosed with a disease, but they have risk factors for illness and have tendency to develop diseases. The term refers to an existing condition of ill health that could lead to a pathologic condition but could also be eliminated, enabling the individual in question to return to a state of good health. Traditional Chinese medicine (TCM) emphasizes the importance of health care and the idea that preventive treatment for diseases is superior to curative treatment. Therefore, early TCM-based intervention can improve the health status of people with SHS. People with SHS often experience such nonspecific symptoms as fatigue; such symptoms are typical of SHS from the perspective of TCM. The present study investigated people with SHS and fatigue as their primary symptom. All enrolled participants completed a physical questionnaire, after which their physiological parameters were monitored using a cloud physiological signal monitoring system to investigate correlations with TCM patterns. Methods: The participants first completed a body constitution questionnaire, the WHO Quality of Life questionnaire, the SHSQ-25 questionnaire, the Epworth Sleepiness Scale, and the Pittsburgh Sleep Quality Index, and subsequently underwent sphygmography to determine their pulse patterns. Analyses of pulse waves were presented in relation to the spectral energy ratio (SER), and SER10 scores represented subtle changes in internal organ blood flow; 13-50-Hz spectrum analysis for pulse delineated any flow energy deviation in organs.

ELIGIBILITY:
Inclusion Criteria:

* Fatigue combined with one or more of the following symptoms of insomnia and higher dreaming frequency, irritability and short temperedness, forgetfulness, chest tightness, lack of concentration, or loss of memory (assessed using the Suboptimal Health Status Questionnaire-25 [SHSQ-25]).
* Body mass index (BMI) between 25 and 30 kg/m2.
* Resting blood pressure measured as 130-139/80-89 mmHg on more than three occasions in 1 week.
* SHSQ-25 score of ≧35

Exclusion Criteria:

* Individuals diagnosed as having a chronic condition by Western medicine, including hypertension, diabetes, chronic hepatitis, chronic kidney disease, chronic hyperlipidemia, and coronary heart disease.
* Individuals diagnosed as having a mental illness by Western medicine.
* Individuals diagnosed with cancer.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study enrolled individuals aged between 20 and 39 years based on previous studies, which showed that SHS is most prevalent in people aged 20 to 39 years. Individuals who conformed to A+B+D or A+C+D (described below) and who had not been diagnosed as having a disease by personnel practicing Western medicine were defined as having SHS. Individuals who did not meet the criteria for SHS and who had not been diagnosed as having a disease by Western medicine were defined as healthy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Sub-optimal Health Status Questionnaire-25 | immediately after interview
  minimum (0) and maximum (100) values; score more than 35 is defined as sub-optimal health

SECONDARY OUTCOMES:
heart rate variability | immediately after interview
  a non-invasive method to evaluate autonomic nervous activity in human

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang-Ming university, Taipei, Taiwan